CLINICAL TRIAL: NCT00956722
Title: Hyperimmune Bovine Colostrum - TRAVELAN™ for Patients With Chronic Hepatitis C Virus Infection Not Responding to Standard Therapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Grant Rawling, Immuron Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Immuron Travelan HCV
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2011-06

CONDITIONS: Asymptomatic Chronic HCV Carriers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Active treatment with Bovine colostrum
  Interventions: Drug: Bovine Colostrum Powder

INTERVENTIONS:
Drug: Bovine Colostrum Powder — Bovine Colostrum Powder (Biogard)

SUMMARY:
This is an exploratory trial of Bovine Colostrum powder to decrease translocation of gut-derived microbial products and immune activation in HCV infection.

The study is designed as a single-arm, open-label, before-and after exploratory trial of 10 weeks of Bovine Colostrum Powder (BCP) to reduce translocation of intestinal microbial products and immune activation in patients suffering from chronic hepatitis C virus (HCV) infection.

The study population will include HCV-infected (genotype 1) men and women, ≥ 18 years of age, not receiving anti-viral therapy at the time of enrollment and for at least the previous 3 months. Having failed previous anti-viral therapy (non responders), HCV recurrence after 72 weeks of therapy, developed side effects which mandated stopping anti viral therapy, or not considered eligible for initiation of such treatment, with a plasma HCV RNA level ≥ 1000 I.U.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection (genotype 1), as documented by a positive anti HCV titer, and confirmed by positive HCV RNA.
* Non responder to previous antiviral therapy, HCV recurrence after 72 weeks of therapy, previous antiviral therapy stopped due to side effects, or not a candidate for treatment with interferon + ribavirin.
* No antiviral therapy for at least 3 months.
* HCV RNA ≥1,000 IU obtained within 30 days prior to study entry.
* Not currently listed for liver transplantation
* Female study subjects of reproductive potential (defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or have not undergone a sterilization procedure (hysterectomy or bilateral oophorectomy) must have a negative serum or urine pregnancy test performed within 48 hours before initiating the protocol-specified medication(s) unless otherwise specified by product labeling.
* All study subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization).
* If participating in sexual activity that could lead to pregnancy, the study volunteer must agree that two reliable methods of contraception will be used simultaneously while receiving the protocol-specified medication and for 1 month after stopping the medication. NOTE: Hormonal-based methods alone are not sufficient. At least two of the following methods MUST be used appropriately unless documentation of menopause, sterilization, or azoospermia is present:

  * Condoms (male or female) with or without a spermicidal agent. Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV transmission;
  * Diaphragm or cervical cap with spermicide;
  * IUD;
  * Hormonal-based contraception.
* Study subjects who are not of reproductive potential (girls who have not reached menarche or women who have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy and/or bilateral oophorectomy are eligible without requiring the use of contraceptives. Written or oral documentation communicated by clinician or clinician's staff is required by one of the following:

  * Physician report/letter;
  * Operative report or other source documentation in the patient record (a laboratory report of azoospermia is required to document successful vasectomy);
  * Discharge summary;
  * Laboratory report of azoospermia;
  * FSH measurement elevated into the menopausal range as established by the reporting laboratory.
* Men and women age > 18 years.
* Ability and willingness of subject or legal guardian/representative to provide informed consent.

Exclusion Criteria:

* Pregnancy or Breast-Feeding
* Continuous use of the following medications for more than 3 days within 30 days of study entry:

  * Immunosuppressives;
  * Immune modulators;
  * Systemic glucocorticoids;
  * Anti-neoplastic agents;
  * Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
To determine if the administration of BCP will reduce the levels of intestinal microbial products in the bloodstream of HCV-infected, untreated persons. | 10 weeks
To determine the safety of the administration of oral BCP to patients with chronic HCV | 12 weeks

SECONDARY OUTCOMES:
To determine whether the administration of BCP will reduce HCV RNA levels or the frequency of T cells expressing markers of cellular immune activation in the peripheral blood of HCV-infected, untreated persons. | 10 weeks
To determine whether the changes in levels of intestinal microbial products in plasma after administration of BCP are associated with changes in HCV RNA levels or the frequency of activated T cells in the peripheral blood | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gadi Lalazar, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Liver Unit, Hadassah Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Brenchley JM, Price DA, Schacker TW, Asher TE, Silvestri G, Rao S, Kazzaz Z, Bornstein E, Lambotte O, Altmann D, Blazar BR, Rodriguez B, Teixeira-Johnson L, Landay A, Martin JN, Hecht FM, Picker LJ, Lederman MM, Deeks SG, Douek DC. Microbial translocation is a cause of systemic immune activation in chronic HIV infection. Nat Med. 2006 Dec;12(12):1365-71. doi: 10.1038/nm1511. Epub 2006 Nov 19. PMID 17115046